CLINICAL TRIAL: NCT04228588
Title: A Pragmatic Study to Investigate the Efficacy and Safety of Mepolizumab in Severe Uncontrolled Asthma in Brazil
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDC 4863/19/082; ISS 212936 (Other Grant/Funding Number: GSK)
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Eosinophilic Asthma
Keywords: severe asthma; mepolizumab; anti IL-5 monoclonal antibody; pragmatic study
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: Phase IV, single-arm study Number of visits: 13 (W-4, W0, W4, W8, W12, W16, W20, W24, W28, W32, W36, W40, W44, W48) (W = week)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mepolizumab (Experimental): Mepolizumab 100mg, SC, every 4 weeks
  Interventions: Drug: Mepolizumab 100 MG [Nucala]

INTERVENTIONS:
Drug: Mepolizumab 100 MG [Nucala] — Mepolizumab 100mg, SC, every 4 weeks

SUMMARY:
The anti-interleukin-5 monoclonal antibody mepolizumab is approved as an add-on therapy in Europe, Canada, USA, and other countries, to standard of care for the treatment of patients with severe eosinophilic asthma. Mepolizumab has been shown to reduce exacerbation rates and dependency on oral corticosteroid use in clinical trials in patients with severe eosinophilic asthma compared with placebo, both in addition to standard of care. Other trials had also showed that treatment with mepolizumab resulted in significant improvements in quality of life (SGRQ) and asthma control (ACQ-5 score) . Mepolizumab has only recently been approved in Brazil. There is still no data regarding its efficacy and safety in the Brazilian population and it is important to emphasize that no Brazilian center participated in the previous large, international and multicentric phase III mepolizumab studies. Therefore, it is crucial to perform a local study in order to validate external results in the Brazilian population.

DETAILED DESCRIPTION:
Severe asthma is associated with substantial morbidity, mortality, health-care costs, and impaired quality of life. Recurrent asthma exacerbations are a major problem in some patients and can predominate in a subgroup with eosinophilic airway inflammation. Mepolizumab is a humanised monoclonal antibody against interleukin 5 that effectively inhibits eosinophilic airway inflammation.

The anti-interleukin-5 monoclonal antibody mepolizumab is approved as an add-on therapy in Europe, Canada, USA, and other countries, to standard of care for the treatment of patients with severe eosinophilic asthma. Mepolizumab has been shown to reduce exacerbation rates and dependency on oral corticosteroid use in clinical trials in patients with severe eosinophilic asthma compared with placebo, both in addition to standard of care. Other trials had also showed that treatment with mepolizumab resulted in significant improvements in quality of life (SGRQ) and asthma control (ACQ-5 score).

Mepolizumab has only recently been approved in Brazil. There is still no data regarding its efficacy and safety in the Brazilian population and it is important to emphasize that no Brazilian center participated in the previous large, international and multicentric phase III mepolizumab studies. Therefore, it is crucial to perform a local study in order to validate external results in the Brazilian population.

Our group belongs to a public academic institution with a focus on assistance, teaching and research. It is a tertiary-referral hospital with an outpatient clinic specializing severe asthma patients. In 2012, the investigators published the first study with the clinical characterization of their cohort of severe asthma and its respective phenotypes. Since then, the investigators have carried out several studies in order to identify prognostic factors and interventions that could improve the control and quality of life of this population. Among them, there are the impact of weight control in asthma symptoms, evaluation of standardized and systematic protocol based on high doses of inhaled corticosteroid plus LABA and 2 weeks course of oral corticosteroids and pathophysiological studies based on bronchial biopsy samples from patients with severe asthma. Since obesity is a serious and prevalent problem in several severe asthma cohorts, another area of interest of the group is to assess the impact of physical activity on this population. Finally, it is important to mention the commitment of the group to evaluate the incorporation of new treatments in the severe asthma population within the Brazilian scenario as done in a specific publication to systematically evaluate the use of omalizumab in our center.

Therefore, the investigators consider that our center has full capacity to conduct a systematic evaluation study of the use of mepolizumab in the population of severe asthma. The investigators aimed to examine the effects of mepolizumab on quality of life, lung function, asthma symptoms and exacerbation rate in patients with severe eosinophilic asthma in a tertiary reference center in Brazil based on real world data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with severe eosinophilic asthma
* Regular use of high-dose inhaled corticosteroids plus other controller medicines
* Non-controlled asthma characterized by ACQ-5 > 1.5 OR chronic oral corticosteroids asthmatic patients (Prednisone 5mg or more for at least 3 months) even if ACQ-5 < 1.5
* History of at least one exacerbation requiring treatment with systemic corticosteroids in the previous 12 months before screening OR chronic oral corticosteroids asthmatic patients (Prednisone 5mg or more for at least 3 months) even without exacerbations
* Blood eosinophil count of at least 300 cells per μL within the 12 months before screening OR a blood eosinophil count of at least 150 cells per μL at screening

Exclusion Criteria:

* Current smokers or former smokers with a history of at least ten pack-years
* Individuals with a concurrent respiratory disease
* Those who had received omalizumab within 30 days before screening
* Patients with severe or clinically significant cardiovascular disease, or other eosinophilic diseases.
* Patients with asthma exacerbation 4 weeks before screening for the study
* Patients with parasitic infection in the 6 months before study entry.
* Patients with substantial uncontrolled comorbidity, possibility of pregnancy
* Patients with history of poor treatment adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-01-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in total score of Saint George's Respiratory Questionnaire (SGRQ) between Week 0 and Week 48 | 48 weeks
  This scales varies from 0 to 100. Higher values means worse quality of life.

SECONDARY OUTCOMES:
Change in the number of clinically significant exacerbations of asthma as defined by: worsening of asthma which requires use of systemic corticosteroids* and/or hospitalisation and/or Emergency Department (ED) visits. | 48 weeks
  significant exacerbations are definied as those requiring at least 3 days of systemic corticosteroids
Change in lung function (Forced expiratory volume in first second - FEV1) | 48 weeks
  Measured by spirometry
Change of asthma control measured by Asthma control questionnaire (ACQ) 5 | 48 weeks
  ACQ varies from 0 to 5 with higher values meaning worse asthma control.
Safety measured by the number of adverse events | 48 weeks
  number of all adverse events
Change of asthma control measured by Asthma Control Test (ACT) | 48 weeks
  ACT varies from 5 to 25 with higher values meaning better asthma control.

OTHER OUTCOMES:
Change of small airway involvement measured by forced oscillometry technique (R5-R20) | 48 weeks
  Measured by forced oscillometry technique
Change of quality of life measured by Asthma Quality of Life Questionnaire (AQLQ) | 48 weeks
  Scores range 1-7, with higher scores indicating better quality of life.
Change of airway inflammation measured by fraction of exhaled nitric oxide (FeNO) | 48 weeks
  Higher levels of FeNO means higher inflammation in the airways
Change of airway inflammation measured by percentage of eosinophils in induced sputum | 48 weeks
  Higher values of sputum eosinophils means higher inflammation in the airways

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Athanazio, MD, PhD, Principal Investigator — Medical Assistant
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No